CLINICAL TRIAL: NCT02133222
Title: Circulating Cell-free DNA in Metastatic Melanoma Patient: Mutational Analyses in Consecutive Measurement Before and After Chemotherapy.
Acronym: AMMAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 13-AOI-04
Record Dates: First submitted 2014-04-30; First posted 2014-05-07 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-03

CONDITIONS: Metastatic (Stage IV) Melanoma
MeSH Terms: conditions — Neoplasm Metastasis; Melanoma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metastatic (stage IV) melanoma (Experimental)
  Interventions: Procedure: blood sample

INTERVENTIONS:
Procedure: blood sample

SUMMARY:
Therapies that target specific molecules markedly inhibit cancer growth in several malignancies, and provide valuable strategies for the treatment of advanced melanoma. In recent years, BRAF and KIT have become established therapeutic targets in melanoma patients showing activating mutations in these oncogenes. However, it is crucial that genetic mutations present in the melanoma lesions are identified if the investigators are to design tailormade therapies for individual patients. The tumour genotypes that determine the selection of molecular-targeted therapies are usually identified in primary tumours; however, primary tumours are not always representative of metastases. Circulating free DNA may be a source of valuable information because it can be obtained via routine blood sampling, it provides real-time information about a patient's current disease state, and it allows monitoring and molecular characterization before and after chemotherapy. The aim of the study is to determine the mutational status in circulating DNA in melanoma metastatic patients, with the Sequenom Mass Array, a next generation sequencing technology. Results obtained before and after treatment will be compared with the primary tumor genotype.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Surgical biopsy for histologic diagnostic
* All melanoma subtypes
* Known genotype BRAF V600
* Affiliation social security
* Consent form signed

Exclusion Criteria:

* Patient with histories of cancer or the other synchronous cancer
* Pregnant women
* Breast-feeding women
* Vulnerable patients: major under guardianship; patient deprived of its rights

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Response to treatment (MRI, Scanner) | at three months
  Comparison between first day and third months

CONTACTS AND LOCATIONS:
Overall Officials: Elodie LONG-MIRA, PH, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France